CLINICAL TRIAL: NCT06063616
Title: The Effect of Reiki Application on Pain Severity and Quality of Life in Patients Receiving Hemodialysis Treatment: Qualitative and Double-blind Randomized Controlled Trial
Brief Title: The Effect of Reiki Application on Pain Severity and Quality of Life in Patients Receiving Hemodialysis Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sultan ÇEÇEN (Other)
Responsible Party: Sponsor-Investigator, Sultan ÇEÇEN, Lecturer, Mersin University
Organization: Mersin University (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: Reiki
Record Dates: First submitted 2023-09-12; First posted 2023-10-02 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2022-03

CONDITIONS: Hemodialysis
Keywords: Hemodialysis; Reiki; Pain; Quality of life; Nursing
MeSH Terms: conditions — Pain | interventions — Therapeutic Touch

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The two interviewers responsible for data collection and the patients were blinded as to which group they were in.
  According to the lists created after block randomization in the computer environment, the researcher and the sham Reiki practitioner evaluated the individuals in the groups in which they would apply and received written consent from those who agreed to participate in the research. It was stated that Reiki treatment would be applied to the patients in both groups and the patients were blinded. The group of patients who agreed to participate in the study was not written on the data collection forms until the end of the study. In addition, the interviewer who collected the data was blinded by ensuring that he did not enter the HD hall before the applications were completed.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Reiki group (Experimental): Level I Reiki was applied to 9 points and nearby areas for 30 minutes, three sessions a week, for a total of four weeks, in the first three hours of the HD treatment, by the researcher who completed his second level training according to the Usui method, in line with the Reiki/Sham Reiki Application Protocol.
  Interventions: Other: Reiki
- Sham Reiki group (Sham Comparator): Sham Reiki was applied to 9 points and nearby areas in accordance with the Reiki/Sham Reiki Application Protocol, for a total of four weeks, three sessions per week, for 30 minutes, in the first three hours of the HD treatment, by two students who had not received Reiki training, and were given training on the application by the researcher.
  Interventions: Other: Sham Reiki

INTERVENTIONS:
Other: Reiki — Level I Reiki was applied to 9 points and nearby areas for 30 minutes, three sessions a week, for a total of four weeks, in the first three hours of the HD treatment, by the researcher, who completed his second level training according to the Usui method, in line with the Reiki/Sham Reiki Application Protocol.
  Arms: Reiki group
Other: Sham Reiki — Sham Reiki was applied to 9 points and nearby areas in accordance with the Reiki/Sham Reiki Application Protocol, for a total of four weeks, three sessions per week, for 30 minutes, in the first three hours of the HD treatment, by two students who had not received Reiki training, and were given training on the application by the researcher.
  Arms: Sham Reiki group

SUMMARY:
Purpose The purpose of this study is to determine the effect of Reiki on pain intensity and quality of life in patients receiving hemodialysis treatment.

Materials and methods The research was conducted as a qualitative study using pretest-posttest, double-blind, randomized controlled study and semi-structured in-depth interview. In this study, patients receiving HD treatment in three separate private dialysis centers in Turkey were randomized to Reiki and sham Reiki groups. In the first three hours of the HD session, in the first three hours of the HD session, three sessions a week for a total of 12 sessions for 30 minutes (min), the first level is applied to 9 main points (crown, forehead, throat, heart, solar plexus, sacral and root chakras, knees, ankles and feet). While applying Reiki, the sham Reiki group was touched at the same points for the same period of time by the uninitiated practitioner. At the beginning and end of the study, Kidney Disease Quality of Life (KDQOLTM-36) scores, Visual Analogue Scale (VAS-Pain) before and after the application, and psychodynamic reactions experienced during the Reiki application after the application were evaluated. At the end of the research, the Reiki group's opinions about the Reiki experience were collected using a form consisting of semi-structured questions.

DETAILED DESCRIPTION:
The fifth stage of chronic kidney disease is called end-stage renal disease (ESRD) and hemodialysis (HD) is offered to patients as a renal replacement treatment option unless a successful kidney transplantation occurs at this stage. Although HD treatment is a treatment option that aims to reduce mortality and morbidity rates and improve the quality of life, it is actually a form of treatment that brings with it different problems. Patients receiving HD treatment experience many physical and psychological symptoms such as pain, fatigue, dyspnea, sleep problems, restless leg syndrome, itching, muscle cramps, nausea-vomiting, loss of appetite, constipation, dry skin, sexual dysfunction, anxiety, depression, and delirium.

In addition, these symptoms bring about social and economic problems and negatively affect the patient's quality of life. In patients with ESRD and receiving HD treatment; The most common symptom is pain due to reasons such as accumulation of fluid and metabolic wastes, comorbid causes such as diabetes, cardiovascular and pulmonary diseases, infections, changes in the musculoskeletal system, HD procedure, carpal tunnel syndrome, and anxiety.

Pharmacological and/or complementary and integrative treatment (TIT) methods are used in the management of pain in patients receiving hemodialysis treatment are used. In pharmacological treatment, analgesics with better metabolic clearance such as fentanyl and hydromorphone are preferred. However, patients' inability to fully express their pain, their unwillingness to increase the already existing medication burden, fear of addiction or side effects of the medications to be used, ethnic or cultural factors, healthcare professionals' inability to evaluate pain adequately and lack of training in pain management are among the reasons for HD patients. There are difficulties in pain management due to reasons such as the lack of a guide on pain management. For this reason, patients prefer TIT methods such as yoga, reflexology, music therapy, relaxation exercises, aromatherapy, acupressure, and Reiki instead of drug treatment.

Reiki, one of the energy-based treatments that has attracted great attention from nurses among TIT methods in recent years; It provides physical, mental and emotional healing by balancing the disrupted energy flow. According to the results of studies conducted on different patient groups; Reiki's vital signs, hemoglobin and hematocrit levels, wound healing, digestive problems, acute and chronic pain, sleep, fatigue, anxiety, fear, depression, stress, relaxation, analgesic use, self-esteem, patient satisfaction, hospital stay, communication, life It has been determined that its quality has positive effects on the side effects of chemotherapy and radiotherapy. However, the results of these studies require careful interpretation due to the limited number of randomized controlled studies, lack of sham and control groups, insufficient sample sizes, differences in population characteristics and protocol, frequency and duration.

While only two studies examining the effect of Reiki on pain in patients receiving HD treatment have been found in the literature, no studies investigating its effect on quality of life have been found. Reiki is a method that can be easily learned, is non-invasive, does not require special equipment, is cost-free, easy to apply, reduces the use of analgesics and has no side effects. In addition, since it increases the quality of life by reducing the severity of pain when applied together with standard treatment, it stands out as one of the different approaches that nurses, especially those who have been with the patient for a long time, can offer to the patient in providing pain management. Based on this point, this study aimed to determine the effect of first-level Reiki, which is applied for a total of 12 sessions for 30 minutes three times a week, in the first three hours of HD, on pain intensity and quality of life in individuals receiving HD treatment.

ELIGIBILITY:
Inclusion Criteria:

* Those who are 18 years of age and over,
* Able to speak Turkish and have no communication problems,
* Receiving HD treatment three times a week for 6 months or longer,
* Without a pacemaker,
* Pain intensity of 4 or more based on the average of two VAS-Pain measurement values evaluated one week apart,
* Having lower extremity pain,
* Does not have any psychiatric disorder,
* Patients over the age of 65 with a Standardized Mini Mental Test (SMMT) score of 24 points and above were included.

Exclusion Criteria:

* Those who are under 18 years of age,
* Having hearing problems,
* Those who do not speak Turkish and cannot communicate,
* Having a pacemaker installed,
* Pain intensity of 3 or less according to the average of two VAS-Pain measurement values evaluated one week apart,
* No lower extremity pain,
* Having any psychiatric disorder,
* Those who have previously received energy-based therapies such as Reiki/therapeutic touch/healing touch,
* Patients over the age of 65 with an SMMT value below 24 were not included in the study.

Ages: 26 Years to 82 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Actual)
Dates: Start 2022-06-06 (Actual); Primary Completion 2022-07-04 (Actual); Study Completion 2022-09-08 (Actual)

PRIMARY OUTCOMES:
Pain severity measurement | Day 1
  "Visual Analog Scale (VAS-Pain)" was applied to the patients in the Reiki and sham Reiki groups before and after application. In VAS-Pain, 1-3 cm is considered a "mild pain" score, 4-6 cm is considered a "moderate pain" score, and 7-10 cm is considered a "severe pain" score.
Initial quality of life measurement | Day 1
  Initial quality of life measurement, "Kidney Disease Quality of Life -KDQOLTM-36" were applied to the patients in the Reiki and sham Reiki groups. Scores in each subscale of the KDQOLTM-36 scale range from 0 to 100, with higher scores indicating better health-related quality of life.

SECONDARY OUTCOMES:
Pain severity measurement at the end of the 12th session | 4 weeks later
  "Visual Analog Scale (VAS-Pain)" was applied to the patients in the Reiki and sham Reiki groups before and after application. In VAS-Pain, 1-3 cm is considered a "mild pain" score, 4-6 cm is considered a "moderate pain" score, and 7-10 cm is considered a "severe pain" score.
Quality of life measurement at the end of the 12th session | 4 weeks later
  Quality of life measurement at the end of the 12th session, "Kidney Disease Quality of Life -KDQOLTM-36" were applied to the patients in the Reiki and sham Reiki groups. Scores in each subscale of the KDQOLTM-36 scale range from 0 to 100, with higher scores indicating better health-related quality of life.

CONTACTS AND LOCATIONS:
Locations (1):
- Sultan Çeçen, Çorum, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
De-identified individual participation data will be made available for all outcome measures.
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code

REFERENCES:
- [Background] Zins S, Hooke MC, Gross CR. Reiki for Pain During Hemodialysis: A Feasibility and Instrument Evaluation Study. J Holist Nurs. 2019 Jun;37(2):148-162. doi: 10.1177/0898010118797195. Epub 2018 Aug 31. PMID 30170509